CLINICAL TRIAL: NCT00116597
Title: Active Specific Intranodal Immunotherapy With a Recombinant Vaccinia Virus Expressing Three Melanoma Associated Epitopes and Two Costimulatory Molecules, Followed by Immunization With Synthetic Melanoma Associated Epitopes. A Phase I/II Trial in Patients With Stages IIb to IV Melanoma
Brief Title: Active Specific Intranodal Immunotherapy of Recombinant Vaccinia Virus in Locally Advanced to Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Michel Adamina, M.D., P.D., M.Sc., University Hospital Basel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT1999017/05.050; SNF grant NPF 37 4037-55151
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Melanoma
Keywords: Active Specific Immunotherapy; Intranodal; Cancer; Melanoma stages IIb to IV; Gene Therapy; Recombinant Vaccinia virus; HLA-A2; Mart-1/Melan-A, Gp-100, tyrosinase; Clinical Trial; Phase I/II
MeSH Terms: conditions — Melanoma; Neoplasms; Vaccinia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: Intranodal immunization with a recombinant vaccinia virus expressing 5 transgenes
Biological: Intranodal booster immunizations with synthetic melanoma associated epitopes

SUMMARY:
The purpose of this study is to assess intranodal immunotherapy in locally advanced to metastatic melanoma patients (American Joint Committee on Cancer [AJCC] stages IIb to IV).

For this, the investigators capitalize on their previous melanoma clinical trial (published by Zajac P et al in Human Gene Ther 2003) and take advantage of a proprietary recombinant vaccinia virus (replication inactivated) expressing 5 minigenes: 3 melanoma associated antigens and 2 costimulatory molecules. Immunization with the recombinant vaccinia virus is followed by 3 boosts with soluble, synthetic melanoma associated antigens.

The patients are immunized intranodally (groin lymph node) under ultrasonographic guidance in an outpatient clinic. The protocol foresees 2 cycles of immunotherapy for alternate weeks and lasts 15 weeks.

DETAILED DESCRIPTION:
The investigators have conducted a phase I/II clinical trial based on the intradermal administration to stage III/IV melanoma patients of a recombinant vaccinia virus encoding tumor associated antigens and costimulatory epitopes for the priming of immune responses, followed by boosts with corresponding synthetic peptides (Zajac P et al in Human Gene Ther 2003). Specific cytotoxic T cells could be induced in a majority of patients following priming, but sustained responsiveness could not be maintained by peptide boosting on a long term basis. Emerging evidence supports the notion that expansion of specific T cells requires trafficking of antigen presenting cells loaded with specific determinants to lymphatic nodes, as induced, among others, by pro-inflammatory stimuli. Therefore, we now adopt the intranodal injection of the immunogenic formulations. As for the former melanoma active specific immunotherapy trial, GM-CSF is used as a supporting cytokine. The epitopes considered are expressed, either all or some of them, in over 90% of the melanomas in Western countries; namely, we immunize with Mart-1/Melan-A epitope 27-35, Gp-100 epitope 280-288 and tyrosinase epitope 1-9. As a consequence, HLA-A2 positivity is mandatory for inclusion in the trial. The 2 costimulatory molecules expressed by cells infected with our replication-incompetent recombinant vaccinia virus are B7.1 (CD80) and B7.2 (CD86).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Histologically proven melanoma in AJCC stages IIb to IV
* Resected, recurrent or disseminated disease
* HLA-A2.1 MHC phenotype
* Karnofsky performance status equal or higher than 70%

Exclusion Criteria:

* Patients younger than 18 years
* Pregnancy or inability to perform anticonception
* MHC phenotype other than HLA-A2.1
* Other concurrent malignant disease
* Estimated life expectancy of less than 6 months
* Allergic skin diseases, including eczema, psoriasis and neurodermitis
* Fever or active infection of the respiratory system
* Concurrent severe cardiac or pulmonary disease (New York Heart Association [NYHA] III and IV)
* Significant impairment of liver or kidney function (bilirubin > 30umol/l, GOT >2.5xN, GPT >2.5xN, alkaline phosphatase >2.5xN, creatinine >1.5xN adapted to the age)
* Impairment of the immune system (leucocyte counts <3000/mm3 or granulocytes counts <1500/mm3)
* Concurrent immunosuppressive therapy
* Preexisting severe anemia (hemoglobin lower than 80 g/l)
* Preexisting thrombocytopenia (platelet counts lower than 75,000/ul)
* Ongoing chemotherapy or chemotherapy completed less than 6 weeks before enrollment in the trial
* Any medical or psychiatric condition which, in the opinion of the treating physician or principal investigator, would unacceptably reduce the safety of the proposed treatment, would impair the delivery of treatment, or would preclude obtaining voluntary informed consent
* Patients receiving any other concurrent investigational treatment, or any other concurrent treatment for their cancer
* Patients who cannot avoid close contact with children less than 3 years of age or with immunocompromised household members

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-11; Primary Completion 2007-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety evaluation
Clinical response
Immune response assessment

SECONDARY OUTCOMES:
Survival (disease-free survival [DFS], overall survival [OS])
Dose adaptation

CONTACTS AND LOCATIONS:
Overall Officials: Michel Adamina, M.D., Principal Investigator — University Hospital, Basel, Switzerland; Daniel Oertli, M.D., Study Chair — University Hospital, Basel, Switzerland; Michael Heberer, M.D., Study Director — University Hospital, Basel, Switzerland; Giulio C Spagnoli, M.D., Principal Investigator — University Hospital, Basel, Switzerland; Walter R Marti, M.D., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Background] Spagnoli GC, Zajac P, Marti WR, Oertli D, Padovan E, Noppen C, Kocher T, Adamina M, Heberer M. Cytotoxic T-cell induction in metastatic melanoma patients undergoing recombinant vaccinia virus-based immuno-gene therapy. Recent Results Cancer Res. 2002;160:195-201. doi: 10.1007/978-3-642-59410-6_23. PMID 12079214
- [Background] Zajac P, Schutz A, Oertli D, Noppen C, Schaefer C, Heberer M, Spagnoli GC, Marti WR. Enhanced generation of cytotoxic T lymphocytes using recombinant vaccinia virus expressing human tumor-associated antigens and B7 costimulatory molecules. Cancer Res. 1998 Oct 15;58(20):4567-71. PMID 9788602
- [Background] Adamina M, Oertli D. Antigen specific active immunotherapy: lessons from the first decade. Swiss Med Wkly. 2005 Apr 16;135(15-16):212-21. doi: 10.4414/smw.2005.10127. PMID 15971113
- [Result] Zajac P, Oertli D, Marti W, Adamina M, Bolli M, Guller U, Noppen C, Padovan E, Schultz-Thater E, Heberer M, Spagnoli G. Phase I/II clinical trial of a nonreplicative vaccinia virus expressing multiple HLA-A0201-restricted tumor-associated epitopes and costimulatory molecules in metastatic melanoma patients. Hum Gene Ther. 2003 Nov 1;14(16):1497-510. doi: 10.1089/104303403322495016. PMID 14577912
- [Result] Oertli D, Marti WR, Zajac P, Noppen C, Kocher T, Padovan E, Adamina M, Schumacher R, Harder F, Heberer M, Spagnoli GC. Rapid induction of specific cytotoxic T lymphocytes against melanoma-associated antigens by a recombinant vaccinia virus vector expressing multiple immunodominant epitopes and costimulatory molecules in vivo. Hum Gene Ther. 2002 Mar 1;13(4):569-75. doi: 10.1089/10430340252809856. PMID 11874634
- [Result] Adamina M, Rosenthal R, Weber WP, Frey DM, Viehl CT, Bolli M, Huegli RW, Jacob AL, Heberer M, Oertli D, Marti W, Spagnoli GC, Zajac P. Intranodal immunization with a vaccinia virus encoding multiple antigenic epitopes and costimulatory molecules in metastatic melanoma. Mol Ther. 2010 Mar;18(3):651-9. doi: 10.1038/mt.2009.275. Epub 2009 Nov 24. PMID 19935776